CLINICAL TRIAL: NCT01550328
Title: Bias Source of Signal in SCOUT DS
Acronym: BSOS
Status: Terminated | Type: Observational
Why Stopped: Protocol no longer meets sponsor objectives
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2721
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes
Keywords: Screening for Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to identify device characteristics, components or subsystems that manifest as screening score bias in SCOUT DS.

DETAILED DESCRIPTION:
In the process of calibrating multiple SCOUT DS units, consistent inter-device score differences were found. These differences could create a bias in the measurement of Diabetes Risk scores (DRS) in human subjects. This study is intended to examine two of the various subsystems of the SCOUT DS to determine whether either of them might be capable of introducing bias into the measurements, with the ultimate aim of eliminating inter-device measurement variation.

The testing of human subjects in this trial is necessary to determine whether variability in the performance of these device subsystems actually affect DRS scores in a real world setting.

The trial will be a prospective, single site, investigational trial. The trial will utilize four SCOUT DS devices. Subjects will report to the investigative site for multiple visits. The number of visits will vary between three to seven visits.

ELIGIBILITY:
Inclusion Criteria:

* Males and/ or females greater than or equal to 18 years of age

Exclusion Criteria:

* Have received investigational treatments in the past 14 days
* Have psychosocial issues that interfere with an ability to follow study procedures
* Are known to be pregnant
* Have scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
* Have been treated in the past month with oral steroid therapy or topical steroids applied to the left forearm. Inhaled steroid therapy is not a basis for exclusion
* Are receiving medications that fluoresce (A list of excluded medications is located in Appendix H)
* Are known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects must be 18 years of age or greater.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine Device Bias | Up to 1 year
  The primary objective of this study is to identify device characteristics, components, or subsystems that manifest as screening score bias in SCOUT DS.
  The study will switch subsystems between devices and if the bias differs by more than 3.5 Diabetes Risk Score units compared to the baseline score, we would conclude that the bias was contained within that particular subsystem

CONTACTS AND LOCATIONS:
Overall Officials: Jon Aase, MD, Principal Investigator — VeraLight, Inc.
Locations (1):
- VeraLight, Albuquerque, New Mexico, United States